CLINICAL TRIAL: NCT03652415
Title: Dry Eye Outcome and Prescription Study
Acronym: DROPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Fight for Sight (Other)
Responsible Party: Sponsor
Other Study IDs: 233506
Record Dates: First submitted 2018-08-23; First posted 2018-08-29 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Dry Eye; Dry Eye Syndrome; Blepharitis; Meibomian Gland Dysfunction; Eye Pain; Punctate Epithelial Keratitis; Punctate Keratitis; Tear Film Insufficiency; Kerato Conjunctivitis Sicca; Eye Diseases
MeSH Terms: conditions — Dry Eye Syndromes; Blepharitis; Meibomian Gland Dysfunction; Eye Pain; Xerophthalmia; Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Artificial tears (classified by MHRA as a medical device) — Use of artificial tears
  Other Names: Lubricant drops or ointment

SUMMARY:
The DRy eye Outcome and Prescription Study (DROPS) is a large observational multicentre study exploring the 'real world' effectiveness of artificial tears in dry eye disease and determinants of efficacy. The aim is to include at least 635 symptomatic dry eye patients who are prescribed artificial tears. All trainees and fellows in London are invited to become collaborators: collaborators are asked to consent patients, assess signs at baseline, and give patients questionnaires at baseline and 4 weeks (for home completion). In tandem, we are conducting a qualitative review of ophthalmologists' prescribing behaviours for dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 years and over) with symptoms* of dry eye disease (with or without signs, with or without blepharitis) who start one or more artificial tears. *Symptoms of dry eye disease include: foreign body sensation, dryness, irritation, itching, burning, stinging or grittiness. When signs are present, symptoms of visual disturbance such as poor vision and blurred vision are sufficient as a symptom of dry eye disease too
* must have best corrected visual acuity in at least one eye of at least 6/12.

Exclusion Criteria:

* lacks capacity (e.g. dementia)
* poor understanding of English
* active other apparent ocular surface disease (including conjunctivitis, abrasion, recurrent erosion syndrome, episcleritis, inflamed pingueculum or pterygium, tumour, infectious keratitis).
* immune ocular pathology (including scleritis and uveitis).
* recent (within the last 3 months) or planned ocular surgery or intravitreal injections.
* current use of other ocular medication, e.g. antiglaucoma drops, g ciclosporine.
* use of artificial tears or ointment in the last 1 month.
* gross lid abnormalities, including significant ectropion or entropion; facial nerve palsy; thyroid eye disease; trichiasis.

For the qualitative interview study:

Subject inclusion criteria

- London NHS Consultant with at least 6 months experience as a Consultant, with a special interest in Cornea and External Diseases, Accident and Emergency and Primary Care, or General Ophthalmology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending hospital ophthalmology outpatient clinics and emergency care (Eye Casualty). Dry eye can be the presenting problem or a secondary problem.
Sampling Method: Non-Probability Sample
Enrollment: 635 (Estimated)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-08-23 (Estimated); Study Completion 2021-08-23 (Estimated)

PRIMARY OUTCOMES:
OSDI | 1 month
  Ocular Surface Disease Index, consists of 12 questions asking about frequency of dry eye symptoms, each scored on a 0-4 scale. Total score varies from 0 to 100, the lower the better. This score is calculated by the sum of the scores for all 12 questions answered multiplied by 100, which is divided by the total number of questions answered times four. It has 3 subscales: vision-related function, ocular symptoms, and environmental triggers, similarly calculated and similarly varying from 0 to 100.
SANDE | 1 month
  Symptom Assessment iN Dry Eye. The two-item SANDE questionnaire score is calculated by multiplying the frequency of symptoms score with the severity of symptoms score and obtaining the square root, leading to a score from 0 to 100. The lower the score, the less severe the symptoms. The answers are given on a 100mm horizontal visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Guys and St Thomas' Hospital, London
  - Guys and St Thomas's Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided